CLINICAL TRIAL: NCT05841758
Title: Hydroxychloroquine as a Steroid-sparing Agent in Extrapulmonary Sarcoidosis: Multicenter, Prospective, Placebo-controlled, Randomized Trial
Brief Title: Hydroxychloroquine as a Steroid-sparing Agent in Extrapulmonary Sarcoidosis
Acronym: CAESAR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL21_1054; 2022-502155-65-00 (Other: EUCT number)
Record Dates: First submitted 2023-03-17; First posted 2023-05-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: Sarcoidosis; Hydroxychloroquine; steroid-sparing agent; Extra pulmonary sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Experimental): prednisone (scheduled protocol) + hydroxychloroquine (200-400 mg /day during a 12 months double blind placebo-controlled period, then according to the treating the physician for an additional open period of 12 months)
  Interventions: Drug: Hydroxychloroquine
- Placebo arm (Placebo Comparator): prednisone (scheduled protocol) + placebo (1-2 tablets/day during a 12 months double blind placebocontrolled period, then the treatment is left to the physician's discretion until M24)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine (200-400 mg /day during a 12 months double blind placebo-controlled period)
  Arms: Hydroxychloroquine
Drug: Placebo — Placebo during a 12 months double blind placebo-controlled period
  Arms: Placebo arm

SUMMARY:
Sarcoidosis is a systemic granulomatous disease of unknown aetiology, mainly affecting the lungs and lymphatics. It affects people worldwide (incidence, 4.7-64/100000; prevalence, 1-36/100000/year). Although it is most often a benign acute or subacute condition, sarcoidosis may progress to a disabling chronic disease in 25% of the cases, with severe complications in about 5%, such as lung fibrosis, cardiac or neurosarcoidosis, defacing lupus pernio or blindness due to uveitis.

When indicated, corticosteroids (CS) are the mainstay of treatment. Due to the kinetics of granuloma resolution, the usual and quite 'dogmatic' duration of treatment is said to be one year, following four classical steps. The long-term use of CS is hindered by cumulative toxicity and efforts have to be made to taper them, as quickly as possible, to the lowest effective dose. A recent report mentioned 39% of the CS-treated patients requiring a steroid-sparing agent. Chloroquine (CQ) and hydroxychloroquine (HCQ) are anti-malarial drugs that have been used since the 1960's as steroidsparing agents on the basis of a landmark study by Siltzbach reporting their efficacy in 43 patients with skin and intrathoracic sarcoidosis. Subsequently, two small randomized controlled trials have shown significant and prolonged improvement on pulmonary symptoms. Only small case series/reports have shown CQ/HCQ efficacy on extra-pulmonary sarcoidosis with response rates ranging from 67 to 100%. Nevertheless, CQ/HCQ are daily used for skin, bone, and joint sarcoidosis, as well as hypercalcemia. Nowadays, HCQ is preferred over CQ because of a lower incidence of gastrointestinal and ocular adverse reactions, which can be minimized by close attention to the dosage and regular retinal examination. Its profile of safety is well-known since it has long been employed to treat systemic lupus erythematous or rheumatoid arthritis. Its action is thought to rely on its ability to accumulate in lysosomes of phagocytic cells, to affect antigen presentation and reduce pro-inflammatory cytokines. The investigator hypothesize that HCQ may be an efficacious add-on therapy for extra-pulmonary sarcoidosis leading to a significant steroid-sparing effect.

ELIGIBILITY:
* Inclusion Criteria :

  * at least 18 years of age
  * pathologically proven sarcoidosis as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)/World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) criteria
  * non severe ocular sarcoidosis requiring systemic treatment
  * non severe skin sarcoidosis requiring systemic treatment
  * non severe osseous sarcoidosis requiring systemic treatment
  * non severe sarcoidosis with joint involvement requiring systemic treatment
  * non severe sarcoidosis-related hypercalcemia requiring systemic treatment
  * non severe peripheral nervous system sarcoidosis requiring systemic treatment
  * non severe sarcoidosis-related non-severe Ear, Nose and Throat (ENT) involvement requiring systemic treatment
  * symptomatic hypercalciuria >200 mg/24h (24 h urine) OR

    * - > 20 mg/mmol creatinine on urine sample
    * - > 180 mg/g creatinine on urine sample
  * signed informed consent
  * affiliated to National French social security system
* Exclusion Criteria :

  * severe sarcoidosis involvement requiring another immunosuppressant or anti-TNF antibody or methylprednisolone i.v. pulses
  * previous (<3 months before screening) or concurrent treatment with immunosuppressants
  * previous treatment with corticoid (patient weaned for 3 months before inclusion)
  * previous treatment with antimalarial drugs (HCQ/CQ) (patient must have been off plaquenil for at least 12 months)
  * treatment with citalopram, escitalopram, hydroxyzin, domperidone and piperaquine
  * known hypersensitivity or intolerance to HCQ/CQ or 4-aminoquinoline derivatives and prednisone
  * heart rhythm disorders on EKG (QT prolongation) (except atrial fibrillations)
  * severe ophthalmological impairment or ophthalmological impairment that does not allow ophthalmic monitoring; previous history of maculopathy or retinopathy
  * end-stage lung, liver, cardiac, or renal disease
  * sarcoidosis with central nervous system involvement
  * cardiac sarcoidosis
  * clinical evidence of active infection (including infection with herpes virus and varicella-zoster virus) or severe/unstabilized comorbidity (e.g. moderate to severe heart failure) or unstabilized psychosis
  * chronic viral (HIV or HBV) infection
  * untreated latent/active tuberculosis
  * pregnancy or lactation (βHCG will be test by blood analysis at inclusion)
  * concurrent vaccination with live vaccines during therapy
  * inability to understand information about the protocol and to sign informed consent or not suitable candidate to comply with the requirements of this study
  * patient participating in other interventional research
  * persons under court protection
  * Use of effective contraception for the duration of the study . (Contraception is considered effective when it consists of one of the following: use of a male condom during all sexual activity and/or efficient oral hormonal contraception (better considered combined contraception) and/or an intrauterine device (IUD) and/or hormone-releasing intrauterine system (IUS) and/or history of bilateral tubal ligation and/or history of vasectomy, provided the male partner is the trial participant's only sexual partner and/or sexual abstinence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the steroid-sparing effect of hydroxychloroquine as an add-on therapy in patients with non severe extra-pulmonary sarcoidosis requiring a systemic treatment. | at Year 1
  The primary endpoint is the percentage of patients in remission and off prednisone at month 9, without relapse until month 12. The primary endpoint will thus be assessed at M12.
  Remission is defined by either complete or partial response. Complete response is defined as the absence of clinical or paraclinical sign of disease activity. Partial response is defined as the persistence of clinical or paraclinical sign of disease activity, which do not require substantial treatment modification (high dose CS, immunosuppressant or anti-Tumor Necrosis Factor (TNF) drugs). Relapse is defined as the persistence, or recurrence of existing manifestations and/or the occurrence of new sarcoidosis manifestations requiring substantial treatment modification.

SECONDARY OUTCOMES:
Organ-specific response assessed by the extra-pulmonary Physician Organ Severity Tool (ePOST) | at Month 0, Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24.
  score comprised between 0 and 6
rate of complete, partial, stable or progression of the disease | at Month 0, Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24.
  Global clinical response will be assessed by the physician as complete, partial, stable, or progression
Assess the total dose of local steroid treatments | at Month 0, Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24.
  Total dose in Gramme of local steroid treatments
Assess the efficacy of HCQ in maintaining the relapse-free survival over a prolonged period | at Month 0, Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24.
  Relapse rate
Assess and compare the eventual reduction of steroid-related toxicity (side effects) | at Month 0, Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24.
  Frequencies of steroid-associated side-effects monitored clinically and biologically
Assess HCQ safety | at Month 3, Month 6 and Month 12
  HCQ safety will be assessed through initial and annual electroretinogram
Assess HCQ safety | at Month 3, Month 6 and Month 12
  HCQ safety will be assessed through initial and annual autofluorescence
Assess HCQ safety | at Month 3, Month 6 and Month 12
  HCQ safety will be assessed through initial and annual electroretinogram or autofluorescence or Optical Coherence Tomography (OCT), yearly eye evaluation and monitoring of eventual Adverse Event (AE)s. An AE will be considered as serious if it leads to HCQ cessation, hospitalization, or death.
Assess HCQ safety | at Month 3, Month 6 and Month 12
  HCQ safety will be assessed through yearly eye evaluation with monitoring of eventual Adverse Event (AE)s. An AE will be considered as serious if it leads to HCQ cessation, hospitalization, or death.
Assess HCQ safety | at Month 3, Month 6 and Month 12
  HCQ safety will be assessed through Optical Coherence Tomography (OCT)
Assess patients' adherence | at Month 3, Month 6 and Month 12
  Patient's adherence will be controlled by patient notebooks
Assess patients' adherence | at Month 3, Month 6 and Month 12
  Patient's adherence will be controlled by pharmacy count of returned tablets
Assess patients' adherence | at Month 3, Month 6 and Month 12
  Patient's adherence will be controlled by serial dosages of blood HCQ levels
Assess quality of life by the Study Short Form 36 questionnaire (SF-36 questionnaire). | at Month 0, Month 1, Month 3, Month 6, Month 12, Month 18 and Month 24.
  11 questions are asked, the minimum score is 36 and the maximum score is 149. Statistical analysis of the SF-36 questionnaire will be performed by a statician, analysis is more complex than only higher score means better health.

CONTACTS AND LOCATIONS:
Locations (21):
- France (21):
  - Service de Médecine Interne Infectiologie Aïgue Polyvalente- Hôpital Henri Duffaud, Avignon
  - Service de Pneumologie - Hôpital Avicenne, Bobigny
  - Service de medecine interne - Hôpital Henri Mondor, Créteil
  - Service de Médecine Interne et Immunologie Clinique - CHU Dijon Bourgogne, Dijon
  - Service de medecine interne - Hôpital Claude Huriez, Lille
  - Service de medecine interne - Hôpital Duputryen, Limoges
  - Service de médecine interne - Hôpital de la Croix Rousse, Lyon
  - Service de médecine interne - Hôpital Edouard Herriot, Lyon
  - Service de médecine interne - Hôpital Lyon Sud, Lyon
  - Service de médecine interne - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Service de medecine interne - Hôpital Saint Eloi, Montpellier
  - Service de medecine interne - Hôpital Hôtel Dieu, Nantes
  - Service de médecine interne - Hôpital Lariboisière, Paris
  - Service de medecine interne 2- Hôpital de la Pitié-Salpétrière, Paris
  - Hôpital Cochin - Médecine interne, Paris
  - Hôpitaux Saint Joseph et Marie LANNELONGUE, Paris
  - Service de Médecine Interne et maladies infectieuses - Hôpital Haut Lévêque, Pessac
  - Service de Médecine Interne et Immunologie Clinique - Hôpital Sud, Rennes
  - Service de medecine interne - Hôpital Nord, Saint-Etienne
  - Service de médecine interne - Clinique Saint exupéry, Toulouse
  - CHU Tours - Médecine interne, Tours

IPD SHARING:
Plan to Share IPD: No